CLINICAL TRIAL: NCT04741919
Title: Randomized Prospective Study of Superior Versus Temporal Laser Peripheral Iridotomy (LPI) in Primary Angle Closure Suspects (PACS)
Brief Title: Superior vs Temporal Laser Peripheral Iridotomy in Primary Angle Closure Suspects (PACS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Catherine Birt, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3236_2020
Record Dates: First submitted 2020-10-16; First posted 2021-02-05 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Primary Angle Glaucoma Closure Suspect

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized to a specific LPI placement (superior or temporal) for one eye, and will be given the other alternative placement for the second eye. This is paired-eye comparative clinical trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superior LPI placement (Active Comparator): Each participant will be randomized to receive an LPI placement superiorly in one eye.
  Interventions: Procedure: Yag Laser peripheral Iridotomy
- Temporal LPI placement (Active Comparator): Each participant will be randomized to receive an LPI placement temporally in one eye.
  Interventions: Procedure: Yag Laser peripheral Iridotomy

INTERVENTIONS:
Procedure: Yag Laser peripheral Iridotomy — Laser peripheral iridotomy will be performed using neo-dynium:yttrium:aluminium-garnet laser after pretreatment with 2% pilocarpine and brimonidine 0.15%. Superior LPIs will be placed between the 11- and 1-o'clock positions such that they were covered completely by the upper eyelid; nasal/temporal LPIs will be placed between the 2- and 4-o'clock positions or the 8- and 10-o'clock positions such that they were completely clear of the lid margin. Preference will be given to iris crypts, avoiding iris vessels when possible. Laser peripheral iridotomies will be performed in both eyes during the same visit and will be confirmed to be patent after the procedure. Intraoperative data collected will include initial per-shot laser energy in milli joules, number of laser shots, and total laser energy in millijoules. All the patients will be treated with flurometholone 0.1% eye drops QID for 5 days after surgery.

SUMMARY:
Basic Study Design: Prospective, randomized, single-center, single-blinded study to compare dysphotopsias and pain recollection immediately 2 weeks, and 3 months after LPI in PACS patients who have a clear indication for bilateral LPI. Our null hypothesis is that there is no difference in dysphotopsia or pain levels by LPI position. Our alternate hypothesis is that there are more dysphotopsias superiorly and more pain temporally.

DETAILED DESCRIPTION:
The study objective is to describe the difference in the incidence of dysphotopsias and sensation of pain both immediately, 2 weeks and 3 months after superior or temporal LPI. The main primary outcome variable will be the presence of dysphotopsias and the recollection of pain graded by a standardized pain scale.

Stratified Block Randomization: 200 patients will be recruited from participating centre. For each patient, the order of the eye to be treated as well as the position of the LPI superior or temporal will be randomized.

Methods:

Subjects: Patients included in the study will be patients referred for a glaucoma evaluation or in follow up at Sunnybrook Science Center who are diagnosed as PACS and have therefore an indication for bilateral LPIs.

Interventions: All patients eligible will be examined by the principal investigator, including a slit lamp assessment of the anterior segment, gonioscopy of the angle and stereoscopic optic nerve examination with a 78 Diopters lens. Intraocular pressure (IOP) will be measured with applanation tonometry. Patients will be assessed with a macular and optic nerve OCT to rule out glaucoma.

Only bilateral PACS patients will be included. One randomly selected eye will receive superior LPI while contralateral eye temporal LPI. At the 2 week and 3 month follow up visits patients will be asked about dysphotopsias in one or both eyes and their recollection of pain will be graded. Other distractors will be included in the questionnaire such as increased tearing sensation.

Laser peripheral iridotomy will be performed using neo-dynium:yttrium:aluminium-garnet laser after pretreatment with 2% pilocarpine and brimonidine 0.15%. Superior LPIs will be placed between the 11- and 1-o'clock positions such that they were covered completely by the upper eyelid; nasal/temporal LPIs will be placed between the 2- and 4-o'clock positions or the 8- and 10-o'clock positions such that they were completely clear of the lid margin. Preference will be given to iris crypts, avoiding iris vessels when possible. Laser peripheral iridotomies will be performed in both eyes during the same visit and will be confirmed to be patent after the procedure. Intraoperative data collected will include initial per-shot laser energy in milli joules, number of laser shots, and total laser energy in millijoules. All the patients will be treated with fluorometholone 0.1% eye drops QID for 5 days after surgery.

Data Collection: Laser treatment specifications will be noted for the amount in LPI positioning, number of applications, and amount of energy used. Other relevant patient information will also be noted such as best corrected visual acuity (BCVA), refractive error, IOP and presence of lens opacities along with the patients gender, age and ethnicity. These patients will be scheduled for follow up examination and IOP measurement at 2 weeks and 3 months after LPI procedure. On follow up a questionnaire will be given to patients assessing pain recollection and presence of dysphotopsias. Lid coverage of the LPI will also be noted.

Sample size and Justification:

The target sample size of 200 participants was selected to provide 80% power on an estimated incidence of 10.7% incidence of dysphotopsias after superior LPI versus 2.4% after temporal LPI with a 2-sided error at α = .05. This was based on the study published by Vera et al,.2014. The sample size allows for a 15% loss to follow-up and a 10% crossover between randomization groups.

Data Analysis: Group differences in baseline variables will be evaluated using Student t test for continuous variables and chi-square tests for categorical variables. P values of less than 0.05 will be considered statistically significant.

Recruitment: Patients will be identified on initial or follow up visits at Sunnybrook Health Center. The ophthalmologists will identify potential subjects and the study coordinator will explain the nature of the study and invite them to participate. An Information and Consent Form will be signed by the patient previous to the enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* clinical evidence of bilateral occludable angles (PACS) defined as:

* Peripheral anterior synechia (PAS) absent and trabecular meshwork not visible in ≥6 clock hours under non-indentation gonioscopy, Along with,
* absence of PAC or PACG, in both eyes.
* macular and optic nerve OCT within the 95% range of the normative database for patients to be included in this study.

Exclusion Criteria:

* evidence of unilateral PACS,
* a history suggestive of an acute angle closure attack (based on symptoms) documented intraocular pressure over 30 mmHg,
* or any sign of Angle Closure Glaucoma (manifest glaucomatous neuropathy detected by OCT).
* Patients with previous ocular surgeries will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dysphotopsias noted from baseline visit before procedure till 3 months after procedure | 3 months from baseline visit
  We will inquire if patients experienced any of the following before and/or after the iridotomy: halo, lines, crescent, ghost image, glare, spots, shadows, blurring, or other unlisted visual disturbances. This will be part of the questionnaire completed before the procedure, at 2 weeks, and at 3 months.

SECONDARY OUTCOMES:
Pain during the baseline visit procedure and recollection of pain till 3 months after procedure | 3 months from baseline visit
  The pain during the procedure and recollection of pain in follow up study visits; (no pain is expected once the procedure is completed) is a secondary outcome, as part of the questionnaire, graded by a standardized pain scale grading the pain from 0 to 10, being 0 no pain and 10 the worst imaginable pain). This will be assessed immediately after the procedure, at 2 weeks and at 3 months after their laser peripheral iridotomy has been performed as is the current standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Birt, MD, FRCSC, Principal Investigator — Sunnybrook
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No